CLINICAL TRIAL: NCT03074864
Title: Intercalated Combination of Erlotinib and Radiotherapy for Patients With EGFR-mutant, Unresectable, Locally Advanced Non-small-cell Lung Cancer
Brief Title: Targeted Treatment With Intercalated Radiotherapy in EGFR-mutant IIIA/IIIB NSCLC
Acronym: TREND
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huajun CHEN, Principal Investigator, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREND
Record Dates: First submitted 2017-02-27; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Non-small Cell Lung Cancer; Epidermal Growth Factor Receptor
Keywords: Activating mutations,lung cancer,radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: EGFR-TKI intercalted with radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EGFR-mutant IIIA/IIIB NSCLC (Experimental): Erlotinib Hydrochloride 150mg daily intercalated with radiotherapy
  Interventions: Drug: Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Subjects receive erlotinib tablet 150mg orally once daily, after 12 weeks of induction phase, local radiotherapy is intercalated, and followed by 24-week erlotinib maintenance phase. At the end of maintenance, the subjects enter into the follow-up period.
  Other Names: Cp-358,774, OSI-774, Tarceva

SUMMARY:
The aim of this study is to investigate the efficacy and safety of intercalated combination of erlotinib and radiotherapy for patients with EGFR-mutant, unresectable, locally advanced NSCLC, and to explore a new treatment strategy for this subset. After Induction by erlotinib, local radiotherapy is intercalated, and followed by 24-week erlotinib maintenance.

DETAILED DESCRIPTION:
Chemoradiation therapy is the standard treatment for unresectable, locally advanced NSCLC, but its efficacy reaches a platform, and treatment-related life threatening toxicity limits its use. The EGFR tyrosine kinase inhibitors (TKIs) produce a dramatic response in patients carrying EGFR activating mutations in the metastatic setting. Multiple prospective trials show that EGFR-TKIs have a better tolerability when compared with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18 years.
2. ECOG performance status 0-2.
3. Pathologically diagnosed of non-small cell lung cancer, and staged as unresectable IIIA/IIIB according the TNM staging system (2009).
4. EGFR activating mutations in exon 18, 19 or 21were detected in tumor tissue or plasma.
5. Measurable disease must be characterized according to RECIST 1.1 criteria.
6. Life expectancy ≥12 weeks.
7. Adequate pulmonary function: FEV1.0 >50% of the normal predicted value, or DLCO >40% of the normal predicted value.
8. Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN); Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3.0 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
9. Adequate renal function: serum creatinine ≤ 1. 5 x ULN, and creatinine clearance ≥ 45 ml/min.
10. Adequate hematological function: Absolute neutrophil count (ANC) ≥1.0 x 109/L, and Platelet count ≥75 x 109/L, and Hemoglobin ≥8 g/dL.
11. Female subjects should not be pregnant or breast-feeding.
12. Written informed consent provided.
13. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Exclusion Criteria:

1. Histologically mixed with small-cell lung cancer.
2. Mutations in EGFR exon 20 are detected.
3. Exposure to prior chest irradiation before the enrollment.
4. Patients with prior chemotherapy or agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
5. History of another malignancy in the last 5 years with the exception of the following: Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted; Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
6. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
7. Existence of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Tumor response will be evaluated through study completion, an average of 6 weeks.
  assessed by the RECIST 1.1 criteria

SECONDARY OUTCOMES:
1 year survival rate | Pts after maintenance phase will receive long-term follow-up including CT scan every 12 weeks for up to 10 years.
  To evaluate the 1 year survival rate of the new strategy.
3 year survival rate | Pts after maintenance phase will receive long-term follow-up including CT scan every 12 weeks for up to 10 years.
  To evaluate the 3 year survival rate of the new strategy.
Progression free survival（PFS） | Occurrence of local or regional progression, distant metastases, or death from any cause from the time of treatment to the occurrence of one of the failure events, whichever occurs first, assessed up to 10 years.
  The product limit estimator developed by Kaplan and Meier will be used.
Overall survival | Time from treatment to death from any cause, assessed up to 10 years.
  The product limit estimator developed by Kaplan and Meier will be used. Their 95% confidence intervals will be estimated.

OTHER OUTCOMES:
Quality of Life (QOL) | Questionnaire of QOL will be recorded for up to 24 weeks.
  To evaluate the Quality of Life (QOL) of subjects during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Jun CHEN, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided